CLINICAL TRIAL: NCT03930147
Title: Monocentric Interventional Study on the Feasibility of the Invasive Mechanical Ventilation Mode "Adaptive Support Ventilation, ASV" in a Pediatric Population and Comparison to Pressure-Control and Pressure-Support Ventilation Modes
Brief Title: Ventilation With ASV Mode in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, FERRY Thomas, Principal Investigator, University of Lausanne Hospitals
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ASV ventilation in children
Record Dates: First submitted 2019-04-12; First posted 2019-04-29 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Mechanical Ventilation
Keywords: Children; Ventilation; Closed-loop mechanical ventilation; Adaptive support ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Two different phases of ventilation (passive versus active) will be monitored in each patient.
  In each phase, two different modes of ventilation will be performed in a randomized order and will be monitored (Pressure-Control Ventilation and ASV during the passive ventilation phase, Pressure-Support Ventilation and ASV during the active ventilation phase). Washout periods will be performed between the different modes of ventilation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Passive phase, Pressure-Control Ventilation / ASV order (Experimental): 90 minutes of Pressure-Control Ventilation, change to ASV mode with 15 to 30 minutes of washout, 90 minutes of ASV. Return to Pressure-Control Ventilation mode at the end of the intervention.
  Interventions: Procedure: ASV ventilation
- Passive phase, ASV / Pressure-Control Ventilation order (Experimental): 90 minutes of ASV, change to Pressure-Control Ventilation mode with 15 to 30 minutes of washout, 90 minutes of Pressure-Control Ventilation.
  Interventions: Procedure: ASV ventilation
- Active phase, Pressure-Support / ASV order (Experimental): 90 minutes of Pressure-Support Ventilation, change to ASV mode with 15 to 30 minutes of washout, 90 minutes of ASV. Return to Pressure-Support Ventilation at the end of the intervention.
  Interventions: Procedure: ASV ventilation
- Active phase, ASV / Pressure-Support order (Experimental): 90 minutes of ASV, change to Pressure-Support Ventilation with 15 to 30 minutes of washout, 90 minutes of Pressure-Support Ventilation.
  Interventions: Procedure: ASV ventilation

INTERVENTIONS:
Procedure: ASV ventilation — Ventilation on ASV mode

SUMMARY:
ASV mode of ventilation is an automatic mode with closed-loop control used for mechanical invasive ventilation in intubated patients. It has been studied in adult patients but not in children.

This interventional physiology study will include 40 children on mechanical invasive ventilation.

DETAILED DESCRIPTION:
The objective of the study is to assess the feasibility of ASV in children and compare physiologic values on ASV mode to Pressure-Control and Pressure-Support mode of ventilation regarding the participant is on active or passive ventilation phase.

Physiologic values will be monitored on different modes of ventilation in a randomized order. Each participant will be his own control regarding the different modes of ventilation. Monitoring will be done during 90 minutes for each mode of ventilation.

Participant will have two different phases of ventilation. The first one is the passive phase (participant does not trigger the ventilator cycle sustainly) in which ASV and Pressure-Control Ventilation will be performed in a randomized order. The second phase will be the active ventilation phase (participant does trigger the ventilator cycle sustainly) in which ASV and Pressure-Support Ventilation will be performed in a randomized order.

ELIGIBILITY:
Inclusion Criteria:

* children on invasive mechanical ventilation admitted in the Pediatric Intensive Care Unit at Lausanne University Hospital
* Body weight > 6kg
* Absence of pulmonary comorbidity
* Age < 10 years

Exclusion Criteria:

* Patient already included in other interventional clinical study
* body weight < 6kg
* age > 10 years
* more than 20% of air leak around endotracheal tube
* chronic or acute pulmonary disease (ARDS, cystic fibrosis, severe asthma, lobectomy, severe bronchomalacia or severe tracheomalacia)
* severe pulmonary hypertension on inhaled nitric oxide treatment
* severe hemodynamic instability (more than 0.5mcg/kg/min of norepinephrine infusion or other high dose vasoactive agent infusion)
* intracranial hypertension (more than 20mmHg if measured) or suspected intracranial hypertension

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Change of respiratory rate | Continuous recording during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Change of tidal volume | Continuous recording during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Change of peak inspiratory pressure | Continuous recording during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation

SECONDARY OUTCOMES:
Evolution of Minute Ventilation | Continuous recording during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Evolution of Mean airway pressure | Continuous recording during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Evolution of inspiratory time | Continuous recording during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Evolution of ratio inspiratory time/expiratory time | Continuous recording during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Evolution of Crs (respiratory system compliance calculated by the ventilator) | Continuous recording during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Evolution of respiratory system resistance | Continuous recording during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Evolution of respiratory system time constant | Continuous recording during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Evolution of positive end expiratory pressure (PEEP) | Continuous recording during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Evolution of the variation of respiratory rate | Continuous recording during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Evolution of the variation of peak inspiratory pressure | Continuous recording during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Evolution of end-tidal CO2 | Continuous recording during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Evolution of the variation of end-tidal CO2 | Continuous recording during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Evolution of transcutaneous CO2 | Recording every 5 minutes during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Evolution of variation of transcutaneous CO2 | Recording every 5 minutes during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Evolution of inspired oxygen fraction | Continuous recording during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Evolution of variation of inspired oxygen fraction | Continuous recording during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Evolution of transcutaneous oxygen saturation | Continuous recording during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Evolution of variation of transcutaneous oxygen saturation | Continuous recording during each monitoring phase of 90 minutes, 360 minutes
  Physiological respiratory value of mechanical ventilation
Evolution of the work load of mechanical ventilation for doctor | monitoring phase of 90 minutes
  Recording of all modification done on ventilator parameters done by doctor during each monitoring phase
Evolution of mechanical ventilation tolerance | monitoring phase of 90 minutes
  Recording of all sedation drugs administered to the participant during each monitoring phase

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ferry, MD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Lausanne University Hospital, Lausanne, Switzerland